CLINICAL TRIAL: NCT04875130
Title: Adrenomedullin in Context With the Diagnose of Pulmonary Embolism and Its Positive / Negative Predictive Value
Brief Title: Adrenomedullin in Context With Pulmonary Embolism
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: PTE/8424-2/2020
Record Dates: First submitted 2021-04-27; First posted 2021-05-06 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism; Adrenomedullin; Biomarker
MeSH Terms: conditions — Pulmonary Embolism | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- confirmed pulmonary embolism: * Patients with intermediate high and high risk of an acute pulmonary embolism with clinical symptoms.
  * On image based procedures confirmed pulmonary embolism (TTE, contrast CT-angiography).
  * Age under 18.
  * Written agreement to the examination.
  Interventions: Diagnostic Test: blood samples

INTERVENTIONS:
Diagnostic Test: blood samples — Taking blood samples (plasma, serum) and measure the level of Adrenomedullin

SUMMARY:
The pulmonary embolism (PE) causes a blockade of the pulmonary arteries typical due to a thrombus which is formed in the lower region of the body or pretty rare to other materials (tumor, air, fat). The working group plans to evaluate the pathology of the thromboembolism in the case of a partial, subtotal or even total pulmonary embolism. The acute PE is still often in the adult population and in many accompanied by death. Etiological the problem occurs through an acute right ventricular failure and leads into severe pulmonal perfusion disorder with shock and hypoxemia. The right diagnose is pretty hard in the clinical day because all symptoms are common and unspecific. To provide the best treatment in short time it is needed to sum up all the symptoms and evaluate the risk of an acute pulmonary embolism and it's morbidity.

The easiest and fastest way treating a PE is to apply a systemic intravenous thrombolysis but bleeding complications are the most common and most frequently side effects. The decision-making process in patients without shock is pretty hard because of having no clear diagnose. Lab parameters and imaging (CT angiography) is important for the best decision in critical ill PE patients but time is sometimes missing.

A possible new biomarker in identifying a PE is adrenomedullin.

Elevated adenomedullin levels in septic patients with left ventricular heart failure, severe dyspnoea and intubated patients are well known, but in the case of PE it wasn't analysed yet. Human adrenomedullin is a protein with 52 amino acid which is produced in the lung and first extracted in the adrenal gland. The sequence homology is pretty similar to the Calcitonin-Gene-Related-Peptide (CGRP)-protein superfamily (vasodilatation). Its precursor is named pro-adrenomedullin peptide and it shows a significant weaker vasodilatation activity compaired to adrenomedullin. Adrenomedullin causes severe hypotonia in scientific studies where it was applied as an intravenous bolus or infusion. This vasodilatation effect concern to the systemic and as well in the pulmonary circulation. Its vasodilatation mechanism is not clarified yet.

The trial is defined as an prospective study, where the investigators would like to measure/analyse the adrenomeulline level in PE patients in the intermediate high and high risk population. The diagnose and treatment of the patients is fixed to the European Society of Cardiology (ESC) recommendations of the cardiology society of 2019 Guidelines on Acute Pulmonary Embolism (Diagnosis and Management of Pulmonary Embolism).

ELIGIBILITY:
Inclusion Criteria:

* Patients with intermediate high and high risk of an acute pulmonary embolism with clinical symptoms.
* On image based procedures confirmed pulmonary embolism (TTE, contrast CT-angiography).
* Written agreement to the examination.

Exclusion Criteria:

* Age under 18.
* Missing written agreement or cancelled agreement on any time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * emergency ward
  * cardial observation ward
  * internal medicine ward
  * intensive care ward
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Is Adrenomedullin (ADM) a useful new biomarker in the diagnose of pulmonary embolism? | admission - 5th day (change in the baseline)
  Measurement: ADM-Kit (ELISA technique) measures the trend level (pg/ml) during observation time.
  - 4 samples are taken

SECONDARY OUTCOMES:
Is it possible to quantify the severity of pulmonary embolism, because of knowing the elevation of adrenomedullin in systemic circulation failure? | through study completion (2 year)
  Comparing CT-angiography imaging, clinical presentation and ADM-level to evaluate correlation between the ADM-level and the severity of the pulmonary embolism.

OTHER OUTCOMES:
Chang of vital parameters (blood pressure) during observation time combined with ADM level. | admission - 5th day (change in the baseline)
  Additionally, the change of vital parameters:
  * blood pressure (mmHg)
  * Mean-Arterial-Pressure (MAP - calculated)
Chang of vital parameters (heart rate) during observation time combined with ADM level. | admission - 5th day (change in the baseline)
  Additionally, the change of vital parameters:
  - pulse (x/min)

CONTACTS AND LOCATIONS:
Overall Officials: Lajos Bogár, MD, Study Chair — University of Pécs - School of Medicine
Locations (2):
- KRAGES - Hospital of Oberwart, Oberwart, Burgenland, Austria
- University Hospital of Pécs, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Voors AA, Kremer D, Geven C, Ter Maaten JM, Struck J, Bergmann A, Pickkers P, Metra M, Mebazaa A, Dungen HD, Butler J. Adrenomedullin in heart failure: pathophysiology and therapeutic application. Eur J Heart Fail. 2019 Feb;21(2):163-171. doi: 10.1002/ejhf.1366. Epub 2018 Dec 28. PMID 30592365
- [Result] Nishikimi T, Nakagawa Y. Adrenomedullin as a Biomarker of Heart Failure. Heart Fail Clin. 2018 Jan;14(1):49-55. doi: 10.1016/j.hfc.2017.08.006. Epub 2017 Oct 7. PMID 29153200
- [Result] Geven C, Kox M, Pickkers P. Adrenomedullin and Adrenomedullin-Targeted Therapy As Treatment Strategies Relevant for Sepsis. Front Immunol. 2018 Feb 19;9:292. doi: 10.3389/fimmu.2018.00292. eCollection 2018. PMID 29520277
- See also: Pulmonary embolism in adults — http://www.uptodate.com/contents/overview-of-acute-pulmonary-embolism-in-adults